CLINICAL TRIAL: NCT01997827
Title: Clinical Performance of Porcelain-fused-to-metal and All-ceramic Resin-bonded Fixed Dental Prostheses in the Anterior Segment - a Randomized Controlled Pilot Study.
Brief Title: Minimal Invasive Rehabilitation of Tooth Loss in the Anterior Segment
Acronym: MIZE-F
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Participants
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Dr. Wolfgang Bömicke, Dr. med. dent., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-083/2013a
Record Dates: First submitted 2013-11-18; First posted 2013-11-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Unsatisfactory or Defective Restoration of Tooth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metal-ceramic RBFDP (Active Comparator): Treatment with a metal-ceramic RBFDP
  Interventions: Device: metal-ceramic RBFDP
- all-ceramic RBFDP (Experimental): Treatment with an all-ceramic RBFDP
  Interventions: Device: all-ceramic RBFDP

INTERVENTIONS:
Device: metal-ceramic RBFDP — Rehabilitation of tooth loss with a metal-ceramic RBFDP
  Arms: metal-ceramic RBFDP
Device: all-ceramic RBFDP — Rehabilitation of tooth loss with an all-ceramic RBFDP
  Arms: all-ceramic RBFDP

SUMMARY:
Tooth loss can be addressed by different rehabilitative strategies. Implant-supported crowns and conventional bridges (fixed dental prostheses [FDPs]) are well established treatment alternatives. Implant therapy is sometimes impossible, however, because of patient-related risk factors or economic issues. In such cases therapy with an FDP requires extensive removal of tooth structure to provide enough space for the restoration and to ensure mechanical retention if the abutment teeth are sound. Alternatives for rehabilitation requiring minor or no preparation of the anchoring teeth are desirable. Resin-bonded bridges meet this demand for minimal invasiveness and have been used clinically successfully. Sometimes, however, patients choose a conventional FDP over a resin-bonded one (RBFDP) for esthetic reasons since the adhesive wings, which are traditionally made of a cobalt-chromium alloy, might be exposed while speaking or smiling or account for a colour change of the abutment teeth. Such patients profit from an all-ceramic RBFDP. Today, the clinical performance of metal-based and all-ceramic RBFDPs has not yet been evaluated under randomized controlled conditions. The aim of this pilot study is to calculate the sample size that allows us to accept the hypothesis that metal- and all-ceramic RBFDPs are similar regarding their clinical performance with adequate statistical power.

ELIGIBILITY:
Inclusion Criteria:

* missing central or lateral incisor
* regular patient of the department of prosthodontics of the university hospital of heidelberg
* willingness to return for recall examinations on a regular basis
* written informed consent
* abutment teeth are vital or sufficiently endodontically treated
* abutment teeth are periodontally stable
* abutment teeth have only little or no defects of the hardsubstances

Exclusion Criteria:

* Pregnancy or breastfeeding
* medically compromised condition not allowing for standard dental treatment
* Patient is not able to give written informed consent
* alcohol or drug abuse
* positive bruxism and parafunctions questionaire
* Bite-Strip > 2
* Attrition Score > 3
* deep bite (Angle class II/2)
* abutment tooth height < 4mm
* untreated symptomatic periodontal or endodontic lesions
* abutment tooth mobility > grade I
* known allergies to materials used in this study
* poor dental hygiene
* planned change of residency

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Success | 12 months
  restoration/abutment teeth without intervention according to the Fédération dentaire internationale (FDI) World dental federation criteria

SECONDARY OUTCOMES:
Color change of the abutment teeth | before tooth preparation, try-in of the framework, 1 week after cementation
  color change measured with a spectrophotometer expressed as ∆E

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Bömicke, Dr. med. dent., Principal Investigator — Department of Prosthodontics, University Hospital Heidelberg, University of Heidelberg
Locations (1):
- Department of Prosthodontics, University Hospital Heidelberg, University of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany